CLINICAL TRIAL: NCT04025177
Title: Pharmacokinetics and Pharmacodynamics of Indomethacin Used for PDA Treatment in Extremely Preterm Neonates <27 Weeks Gestational Age
Brief Title: Indomethacin PK-PD in Extremely Preterm Neonates
Acronym: INDO
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Halted due to feasibility issues
Sponsor: University of Manitoba (Other)
Collaborators: St. Boniface Hospital (Other); Health Sciences Centre, Winnipeg, Manitoba (Other); University at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2018:095
Record Dates: First submitted 2019-05-27; First posted 2019-07-18 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2020-03

CONDITIONS: Patent Ductus Arteriosus After Premature Birth
Keywords: Indomethacin; Pharmacokinetics; Preterm birth; Pharmacodynamics
MeSH Terms: conditions — Premature Birth | interventions — Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neonates with an open PDA (Experimental): Neonates born between 23 (0/7) and 26 (6/7) weeks gestational age with an open PDA, according to clinical protocol criteria, and no contraindication to the use of indomethacin.
  Interventions: Drug: Indomethacin Injection

INTERVENTIONS:
Drug: Indomethacin Injection — The dose of indomethacin will be 0.1 mg/kg/dose, based on birth weight, intravenously every 24 hours for a total of 3 doses. Doses 2 and 3 may be administered between 23.5 and 24.5 hours after the previous dose. Doses will be rounded to two significant figures.

SUMMARY:
This is a phase II open-label study evaluating the pharmacokinetics and pharmacodynamics of targeted early use of indomethacin for PDA treatment in preterm neonates <27 weeks' gestational age.

DETAILED DESCRIPTION:
Neonates will be enrolled following an echocardiogram performed within 12 hours after birth that confirms an open PDA (with no other contraindications for indomethacin treatment). After enrollment, neonates will receive intravenous indomethacin at a dose of 0.1mg/kg every 24 hours for 3 days. Indomethacin levels will be measured at regular intervals. Urine output and serum electrolytes will be monitored prior to each dose of indomethacin. An echocardiogram will be repeated after completion of indomethacin treatment (between 72-120 hours of age) to reassess the status of PDA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female infant born between 23 (0/7) and 26 (6/7) week GA
* Infant diagnosed with PDA according to clinical protocol criteria
* Able to adhere to indomethacin administration protocol
* The patient is born in the study center.
* Subject's parent(s)/legal guardian(s) has provided signed and dated informed consent and authorization to use protected health information, as required by national and local regulations.
* In the investigator's opinion, the subject's parent(s)/legal guardian(s) understand(s) and can comply with protocol requirements, instructions, and protocol-stated restrictions, and is likely to complete the study as planned.

Exclusion Criteria:

* known major congenital malformations (renal, cardiac, gastrointestinal and central nervous system)
* genetic syndromes-inborn errors of metabolism
* severe renal compromise
* intrauterine growth retardation with birth weight <3rd centile
* thrombocytopenia <50,000/mm3
* moderate to severe pulmonary hypertension
* clinical sepsis -meningitis- hepatitis
* anticipated drug-drug-interactions (specifically CYP2C9, CYP2C19 and UGT 1-1)

Ages: 23 Weeks to 26 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Area under the curve from serial Indomethacin levels | At 48 hour following the last dose
  Blood samples will be drawn from patients to determine the serum indomethacin levels to determine the area under the curve

SECONDARY OUTCOMES:
Percentage of Participants with Patent Ductus Arteriosus Closure | Within 48 hrs after the last dose
  Confirmed by echocardiogram
Percentage of Participants with Intraventricular hemorrhage | Within the first 7 days of life.
  Confirmed by cranial ultrasound performed and graded using Papile's classification system
Duration of mechanical ventilation of each patient | trough hospital discharge, an average of up to 36 weeks gestational age
  Number of days the infant was intubated and ventilated.
Percentage of Participants with Adverse Events | trough hospital discharge, an average of up to 36 weeks gestational age
  development of any type A adverse reactions in the infants receiving indomethacin therapy

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Louis, MD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - St. Boniface General Hospital Research Centre, Winnipeg, Manitoba
  - Health Sciences Centre, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No